CLINICAL TRIAL: NCT05997745
Title: Effects of Early Enteral Nutrition With a Locally Produced Protein-energy Ration Versus a Marketed Nutritional Solution in Patients Operated on for Acute Generalized Peritonitis
Brief Title: Enteral Nutrition in Acute Generalized Peritonitis
Acronym: PAG/NUTRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Evangélique enAfrique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 002
Record Dates: First submitted 2023-08-07; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Enteral and Supplement Feeds Adverse Reaction; Peritonitis; Acute
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): an intervention arm consisting of patients who will receive the locally manufactured protein-energy ration after a laparotomy indicated for generalized acute peritonitis
  Interventions: Dietary Supplement: study group
- control group (Active Comparator): patients who will receive the commercially available protein-energy ration after a laparotomy indicated for generalized acute peritonitis
  Interventions: Dietary Supplement: study group

INTERVENTIONS:
Dietary Supplement: study group — Patients will receive early enteral locally nutrition postoperatively following surgery for peritonitis

SUMMARY:
Hospitals in South Kivu always have problems supplying artificial enteral nutritional products because of their high cost and low availability in our areas. While the Province has cereals, knowing their nutritional composition would enable the formulation of a nutritional product based on local protein-energy products. Hence the questions below: Can a local cereal-based protein-energy ration be used instead of a costly imported artificial nutritional solution to improve the nutritional status of patients operated on for PAG? What is the tolerance of this early enteral nutrition on the healing and functional recovery of patients compared with an artificial nutritional solution? To answer these questions, a randomized clinical trial has been designed with the following objectives:

* To formulate an enteral diet using cereals available in our environment with a protein-calorie composition superimposable on the artificial enteral ration,
* Evaluate the tolerance and advantages of early enteral nutrition with a locally manufactured protein-caloric ration vs. a commercially available artificial nutritional solution in patients undergoing surgery for PAG.

ELIGIBILITY:
Inclusion Criteria:

* patient operated for peritonitis with intestinal suture during treatment
* have a q-SOFA score of 1 to 2
* surgeon's agreement to enteral feeding
* at risk of malnutrition (BMC)

Exclusion Criteria:

* q SOFA score > 2
* patients with tare (diabetes, HIV, renal failure)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability of feeding | 10 days after surgery
  We will screen complications after feeding

SECONDARY OUTCOMES:
nutritional surveillance | 2 days after, 5 days after, 10 days after feeding
  changes in nutritional status using body mass index, albumin measurement, anthropometric data